CLINICAL TRIAL: NCT04417036
Title: Safety and Efficacy of Inhaled Pegylated Adrenomedullin (PEG-ADM) in Patients Suffering From Acute Respiratory Distress Syndrome (ARDS): a Double-blind, Randomized, Placebo-controlled, Multicenter Phase 2a/b Clinical Trial
Brief Title: This Study Collects Information on the Safety of Inhaled Pegylated Adrenomedullin (PEG-ADM), How the Drug is Tolerated and How it Affects Patients Suffering From a Type of Lung Failure That Cause Fluid to Build up in the Lungs Making Breathing Difficult (ARDS)
Acronym: SEAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated (based on Part A results, Bayer decided to not continue investigating BAY 1097761 further in Part B; this was not due to any safety data for BAY 1097761)
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19999; 2019-001078-27 (EudraCT Number)
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part A - Active Drug Dose 1 (Experimental): Participants will receive Active Drug Dose 1 for a maximum of 14 days in study phase Part A
  Interventions: Drug: BAY1097761 Active Dose 1
- Part A - Active Drug Dose 2 (Experimental): Participants will receive Active Drug Dose 2 for a maximum of 14 days in study phase Part A
  Interventions: Drug: BAY1097761 Active Dose 2
- Part A - Placebo (Placebo Comparator): Participants will receive Placebo for a maximum of 14 days in study phase Part A
  Interventions: Other: Placebo to BAY1097761
- Part B - Active Drug Dose (Experimental): Participants will receive Active Drug 1 or 2 for a maximum of 14 days in study phase Part B
  Interventions: Drug: BAY1097761 Active Dose 1; Drug: BAY1097761 Active Dose 2
- Part B - Placebo (Placebo Comparator): Participants will receive Placebo for a maximum of 14 days in study phase Part B
  Interventions: Other: Placebo to BAY1097761

INTERVENTIONS:
Drug: BAY1097761 Active Dose 1 — Participants will receive a lower dose ADM by inhalation
  Arms: Part A - Active Drug Dose 1; Part B - Active Drug Dose
Other: Placebo to BAY1097761 — Participants will receive Placebo to BAY1097761 by inhalation
  Arms: Part A - Placebo; Part B - Placebo
Drug: BAY1097761 Active Dose 2 — Participants will receive a higher dose ADM by inhalation
  Arms: Part A - Active Drug Dose 2; Part B - Active Drug Dose

SUMMARY:
The study is composed of two parts. In part A of the study two active doses of inhaled pegylated adrenomedullin (PEG-ADM) will be compared regarding safety and efficacy to a substance that has no therapeutic effect (placebo) in order to find an optimal and safe of the study drug. In part B of the study the highest dose that is considered safe and has demonstrated efficacy will be taken forward to collect information how well patients suffering from Acute Respiratory Distress Syndrome (ARDS) respond to treatment with inhaled pegylated adrenomedullin (PEG-ADM) compared to treatment with placebo. ARDS is a type of lung failure that cause fluid to build up in the lungs making breathing difficult or impossible.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of inclusion into study.
* Invasively mechanically ventilated acute respiratory distress syndrome [ARDS] patients (diagnosed according to Berlin definition of ARDS, including positive end-expiratory pressure [PEEP] of ≥5 cm H2O, X-ray (or CT scan) indicative of ARDS: bilateral opacities not fully explained by cardiac failure, fluid overload, lobar/lung collapse, effusions or nodules).
* Initial diagnosis of mild, moderate or severe ARDS prior to study inclusion, with acute onset of ARDS within 1 week after suspected trigger factor of

  * Pneumonia
  * Aspiration
  * Sepsis
  * Pancreatitis
* Prior to randomization, hypoxemia with PaO2:FiO2 ≤300 mmHg continuously observed for a period of ≥4 hours (with values of ≥2 arterial blood gas [ABG] analyses during that time, with the last value obtained timely (generally ≤3 hours) prior to randomization), under ventilation with minimum PEEP ≥8 cm H2O.
* Time from first meeting the last diagnostic ARDS criterion (Berlin criteria) to randomization must be ≤48 hours.
* For Study Part A: ARDS patients for whom measurements of extra-vascular lung water are regarded as medically indicated by the treating physician, and these measurements are planned as part of their clinical care, from Study Day 1 up to Study Day 7 (if then still intubated).

Exclusion Criteria:

* Any value of a PaO2:FiO2 ratio >300 mmHg within a time interval of 4 hours before randomization
* Rescue therapy (e.g. inhalation of nitric oxide gas and/or inhalation of prostacyclin analogues, or extra corporeal membrane oxygenation [ECMO] / extra corporeal CO2 removal [ECCO2R]) already initiated at screening and/or Study Day 1 (prior to first dose of the study intervention)
* Moribund participants not expected to survive 24 hours (clinical decision)
* Expected duration of invasive mechanical ventilation less than 48 hours (clinical decision)
* History of co-morbidities requiring long-term/home oxygen use (e.g. severe chronic obstructive pulmonary disease [COPD], pulmonary fibrosis) or non-invasive ventilation (except for sleep apnea management), or making weaning per se improbable (e.g. ALS, muscular dystrophy)
* Smoke inhalation injury, extensive burns or trauma/head injury as concomitant condition
* History of pneumectomy, lung lobectomy or lung transplant
* Diffuse alveolar hemorrhage from vasculitis
* Current lung malignancy (incl. lung metastasis), or other malignancy requiring chemotherapy or radiation within the last month
* Chronic kidney disease with a history of renal replacement therapy (e.g. dialysis)
* Chronic liver disease Child-Pugh Class C
* Chronic heart failure NYHA IV
* Known hypersensitivity to polyethyleneglycol (PEG, Macrogol)
* Participation in other interventional studies involving pharmacological interventions, or biological or cell therapy interventions
* Diagnosis of COVID-19 pneumonia within 6 weeks prior to study inclusion. History of SARS-CoV-2 infection (positive test based on nucleic acid amplification technology or positive antigen test) without COVID-19 pneumonia does not exclude patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
VFS in Part B participants | At Day 28
  Ventilator-free survival (VFS, participants alive and not on invasive mechanical ventilation)

SECONDARY OUTCOMES:
CUI in Part A participants | Up to 7 days
  Clinical Utility Index (CUI) is a summary measure used to compare different treatments, the index score will range between 0 and 1.
VFS in Part A participants | At Day 28
  Ventilator-free survival (VFS, participants alive and not on invasive mechanical ventilation)
All-cause mortality in Part A and Part B participants | At Day 28, Day 60 and Day 90
Proportion of participants who still require invasive mechanical ventilation support in Part A and Part B participants | At Day 28 and Day 60
Ventilator-free days (VFDs) in Part A and Part B participants | Within Day 28 and Day 60
VFS in Part A and Part B participants | At Day 60
  Ventilator-free survival (VFS, participants alive and not on invasive mechanical ventilation)
Integrated analysis on VFS invoving all participants from Part A and Part B | At Day 28 and Day 60
  Ventilator-free survival (VFS, participants alive and not on invasive mechanical ventilation)

CONTACTS AND LOCATIONS:
Locations (22):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Universitätsklinikum AKH Wien, Vienna
- Czechia (3):
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
  - Masaryk Hospital Usti n/L, Ústí nad Labem
- France (6):
  - Centre Hospitalier Universitaire - Angers, Angers
  - Center Hospitalier Michallon - Grenoble, La Tronche
  - Hôpital du Nord - Marseille, Marseille
  - Hôpital de la Pitié-Salpétrière, Paris
  - Cochin - Paris, Paris
  - Hôpital Civil - Strasbourg, Strasbourg
- Germany (3):
  - Klinikum Oldenburg AöR, Oldenburg, Lower Saxony
  - Klinikum der Stadt Köln gGmbH - Krankenhaus Merheim, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel, Schleswig-Holstein
- Italy (3):
  - Istituto Clinico Humanitas - Humanitas Mirasole S.p.A., Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - ASST Santi Paolo e Carlo, Milan, Lombardy
- Spain (3):
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
- United Kingdom (2):
  - University Hospital of Wales, Cardiff
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Karagiannidis C, McAuley DF, Thompson BT, Reimer T, Shakery K, Schmitz S, Cortes MN, Ullrich R, Meziani F, Mercat A, Chiumello D, Duska F, Combes A; SEAL Trial Investigators. Safety and efficacy of inhaled PEG-ADM in ARDS patients: a randomised controlled trial. Crit Care. 2025 Oct 23;29(1):448. doi: 10.1186/s13054-025-05617-y. PMID 41131549